CLINICAL TRIAL: NCT05095480
Title: Does Adding Red Yeast Rice to Statin Can Improve Lipid Profile or Vascular Inflammation? A Randomized Clinical Trial
Brief Title: Effect of Red Yeast Rice Beside Statin on Lipid Profile
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Kojuri, Professor, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SUMS.MED.REC.1399.840
Record Dates: First submitted 2021-10-01; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Hyperlipidemias
Keywords: Hyperlipidemia; Statin; Lesstat; Red Yeast Rice
MeSH Terms: conditions — Hyperlipidemias | interventions — red yeast rice

STUDY DESIGN:
Intervention Model Description: treatment and placebo received their drugs in their group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lesstat (Experimental): Those who received Lesstat
  Interventions: Drug: Red Yeast Rice Pill
- Placebo (Placebo Comparator): Those who received Lesstat
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Red Yeast Rice Pill — Taking Lesstat
  Other Names: Lesstat
  Arms: Lesstat
Drug: Placebo — Placebo receiving group
  Arms: Placebo

SUMMARY:
We conducted a triple-blind clinical trial on 92 patients in 2019. They were randomly divided into a control group of 49 patients and a treatment group of 43 patients. Treatment group received Lesstat and placebo group received the same color tablets

DETAILED DESCRIPTION:
A triple-blind clinical trial on 92 patients in 2019 was conducted. Patients were randomly divided into a control group of 49 patients and a treatment group of 43 patients. The block randomization method with a block size=2 and a ratio of 2:2 for drug vs. placebo was used. Participants were selected from cardiology center (Prof. Kojuri cardiology clinic, Niayesh St., Shiraz, Iran, www.kojuriclinic.com, Instagram @Kojuri_clinic) who took part in this trial voluntarily and were completely informed about the study.

Primarily, some blood tests were done for all of the participants in order to measure their serum levels of LDL cholesterol (LDL-C), HDL cholesterol (HDL-C), total cholesterol, triglyceride (TG), and high sensitivity C-reactive protein (hs-CRP). The patients with very high levels of serum LDL-C (above 200 mg/dL) and those with serum levels of LDL-C below 100m/dL were excluded from the trial.

Food supplements based on red yeast rice were given to the patients of the treatment group in the form of tablets named Lesstat® (Gricar chemical Srl Co.). Each tablet contained 200 mg fermented red rice with Monascus Purpureus tit 5% in Monacolin K, 10 mg equal to Monacolin K, 90 mg chitosan, 3.5 mg lycopene, 30 mg ascorbic acid (vitamin C), and 5 mg tocopherol (vitamin E).

In order to ensure blindness, the placebo tablets were similar to Lesstat (RYR) tablets in shape and color. Both RYR and placebo tablets were given to the patients in identical packages and every package contained 30 tablets of RYR or placebo, which was designed for a one-month use.

After the prescription, the participants were told to take one tablet daily in addition to their routine statin therapy for a period of 30 days. The patients were encouraged to contact us if they had any problems during that 30-day period.

All participants were told to come back to our center after one month in order to perform some secondary blood tests to compare patients' serum levels of LDL-C, HDL-C, total cholesterol, TG, and hs-CRP with the initial measures. We carried out both primary and secondary blood tests in the same laboratory and with the use of the same kits. Additionally, the levels of serum glutamic-oxaloacetic transaminase (SGOT), serum glutamic-pyruvic transaminase (SGPT), and serum total bilirubin of all patients were assessed in order to assess possible adverse hepatic effects of this combination (statins and RYR) therapy.

IBM SPSS software (version 25) for statistical analyses was sed. For comparing the variables between the treatment and placebo groups at baseline, the independent sample t-test and Pearson chi-squared test were . The paired-sample t-test and repeated measure ANOVA were used for the variables with repeated measures. Values of p less than 0.05 were considered to be statistically significant.

All of the participants were totally informed about the purposes and details of our study, with giving their informed consent before taking part. Patients refusing to participate were excluded from the trial.

ELIGIBILITY:
Inclusion Criteria:

* Having serum levels of LDL cholesterol (LDL-C) at least 100 mg/dL and being treated with any group of statins for at least 3 months prior to the trial.

Exclusion Criteria:

* Having very high serum levels of LDL-C (above 200 mg/dL)
* Hypersensitivity to orlistat
* Using other lipid-lowering agents with statins
* History of liver disease
* Pregnancy.

Ages: 55 Years to 72 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Total cholesterol level | 1months
  The level of total cholesterol, mg/dl
Rise of SGOT ( AST) | 1 months
  Rise of serum SGOT,(AST) as liver enzyme, unit per liter
HS-CRP | 1 months
  Inflammation of intravascular, and surrogate marker of atherosclerosis activity, pico/dl
LDL level | 1 months
  The serum level of LDL cholesterol, mg/dl
Triglyceride level | 1 months
  The serum level of triglyceride, mg/dl
HDL cholesterol | 1 months
  The serum level of HDL cholesterol, mg/dl
SGPT( ALT) level | 1 months
  The serum level of SGPT( ALT) U/L
CPK | 1 months
  Serum CPK level , IU/L

SECONDARY OUTCOMES:
Muscular pain | 1 months
  Severe muscular pain, based on patient report
GI upset | 1 months
  Any sever gastrointestinal symptoms, reported by patient

CONTACTS AND LOCATIONS:
Overall Officials: javad kojuri, MD, Principal Investigator — Professor Kojuri Cardiology clinic
Locations (1):
- Javad Kojuri, Shiraz, Outside of the US, Iran

IPD SHARING:
Plan to Share IPD: No
only the result of study is available

REFERENCES:
- [Derived] Tavan A, Noroozi S, Zamiri B, Gholchin Vafa R, Rahmani M, Mehdizadeh Parizi M, Ahmadi A, Heydarzade R, Montaseri M, Hosseini SA, Kojuri J. Evaluation the effects of red yeast rice in combination with statin on lipid profile and inflammatory indices; a randomized clinical trial. BMC Nutr. 2022 Nov 25;8(1):138. doi: 10.1186/s40795-022-00639-z. PMID 36434733